CLINICAL TRIAL: NCT00656188
Title: A Randomized, Double-blind, Parallel-group, Placebo-controlled Study Evaluating the Efficacy and Safety of Vardenafil Administered for 12 Weeks in a Flexible-dose Regimen Compared to Placebo in Male Erectile Dysfunction Subjects
Brief Title: Placebo-controlled Study Evaluating the Efficacy and Safety of Vardenafil in Subjects With Erectile Dysfunction
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10898; GSK 001
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Vardenafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 1 (Active Comparator)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — Vardenafil 5mg or 10mg or 20mg taken orally on demand 1 hour prior to sexual intercourse
  Arms: Arm 1
Drug: Placebo — Matching placebo
  Arms: Arm 2

SUMMARY:
This study tested the hypothesis that vardenafil was both clinically effective and well-tolerated compared to placebo in men diagnosed as being unresponsive to sildenafil.

ELIGIBILITY:
Inclusion Criteria:

* Men >/= 18 years of age, with 6 months or longer diagnosis of ED as defined by NIH Consensus statement,
* History of unresponsiveness to sildenafil
* Stable sexual relationship for > 6 month

Exclusion Criteria:

* Primary hypoactive sexual desire
* History of myocardial infarction, stroke or life-threatening arrhythmia within prior 6 month
* Nitrate therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2002-10; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Erectile Function domain of the International Index of Erectile Function | 12 weeks
Sexual Encounter Profile Question 2 | 12 weeks
Sexual Encounter Profile Question 3 | 12 weeks

SECONDARY OUTCOMES:
Erectile Function domain scores > 26 | 12 weeks
Sexual Encounter Profile 2 | 12 weeks
Global Assessment Question | 12 weeks
Reliability of insertion | 12 weeks
Reliability of maintenance | 12 weeks
Other subject diary based variables | 12 weeks
Safety and tolerability | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer